CLINICAL TRIAL: NCT04498390
Title: A Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of LY3493269 in Healthy Participants
Brief Title: A Safety Study of LY3493269 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17451; J1X-MC-GZHB (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3493269 (Experimental): 8, 24 or 48 milligrams (mg) LY3493269 + 250 or 500 mg permeation enhancer sodium caprate(C10) Once daily (QD) administered orally over 3 consecutive study days.
  Interventions: Drug: LY3493269
- Placebo (Placebo Comparator): Placebo administered orally over 3 consecutive study days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3493269 — Administered orally.
  Arms: LY3493269
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main purpose of this study in healthy participants is to learn more about the safety of LY3493269 and any side effects that might be associated with it. Blood tests will be performed to check how much LY3493269 gets into the bloodstream and how long it takes the body to eliminate it. For each participant, the study will last about 10 weeks and may include 12 visits, including five nights in a row in the clinical research center.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female not of childbearing potential
* Body mass index within the range of 19.0 to 40.0 kilograms per square meter (kg/m²) (inclusive)
* Participants who are healthy as determined through medical evaluation including screening medical history, physical examination, vital signs, clinical laboratory tests, and electrocardiogram (ECG)
* Have clinical laboratory test results within normal reference range for the population or clinical research unit (CRU), or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have glycated hemoglobin level of less than (<)6.5 percent (%)

Exclusion Criteria:

* Have a supine heart rate (HR) less than 50 beats per minute (bpm) or greater than 100 bpm. If a repeat measurement shows values within the range, the participant can be included in the trial
* Have a mean supine systolic blood pressure (BP) higher than 160 millimeters of Mercury (mmHg) and a mean supine diastolic BP higher than 95 mmHg from 2 assessments at screening (excluding white-coat hypertension); therefore, if a repeated measurement shows values within the range, the participant can be included in the trial
* Have undergone any form of bariatric surgery
* Have a history of gastrointestinal (GI) bleeding or duodenal ulcers
* Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2
* Have a history of acute or chronic pancreatitis, or elevation in serum lipase and/or amylase levels greater than 1.5 times the upper limit of normal (ULN)
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis
* Have been treated with prescription drugs that promote weight loss within 3 months prior to screening
* Have participated within the past 30 days of screening in a clinical study involving an investigational product (IP); at least 5 half-lives or 30 days, whichever is longer, should have passed
* Have an abnormality in the 12-lead ECG at screening that, in the opinion of the investigator, increases the risks associated with participating in the study or may confound ECG (QT) data analysis, such as a QT interval corrected using Fridericia's formula (QTcF) greater than (>)450 milliseconds (msec) for males and >470 msec for females, short PR interval (<120 msec), or PR interval >220 msec, second and third atrioventricular block, intraventricular conduction delay with QRS >120 msec, right bundle branch block, left bundle branch block or Wolff-Parkinson-White syndrome
* Have serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times (X) ULN or total bilirubin level (TBL) >1.5X ULN
* Have known allergies to LY3493269, related compounds, or any components of the formulation (including C10), or a history of significant atopy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo once daily (QD) administered orally over 3 consecutive study days.
- Cohort 1: 8 Milligrams (mg) LY3493269 + 500 mg C10: Participants received 8 mg LY3493269 + 500 mg permeation enhancer sodium caprate(C10) QD administered orally over 3 consecutive study days.
- Cohort 2: 24 mg LY3493269 + 500 mg C10: Participants received 24 mg LY3493269 + 500 mg C10 QD administered orally over 3 consecutive study days.
- Cohort 3: 48 mg LY3493269 + 500 mg C10: Participants received 48 mg LY3493269 + 500 mg C10 QD administered orally over 3 consecutive study days.
- Cohort 4: 24 mg LY3493269 + 250 mg C10: Participants received 24 mg LY3493269 + 250 mg C10 QD administered orally over 3 consecutive study days.
Period: Overall Study
Arm/Group | Placebo | Cohort 1: 8 Milligrams (mg) LY3493269 + 500 mg C10 | Cohort 2: 24 mg LY3493269 + 500 mg C10 | Cohort 3: 48 mg LY3493269 + 500 mg C10 | Cohort 4: 24 mg LY3493269 + 250 mg C10
Started | 8 | 8 | 8 | 8 | 8
Received at Least One Dose of Study Drug | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 7 | 7 | 8
Not Completed | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Cohort 1: 8 mg LY3493269 + 500 mg C10: Participants received 8 milligrams (mg) LY3493269 + 500 mg permeation enhancer sodium caprate(C10) QD administered orally over 3 consecutive study days.
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort 1: 8 mg LY3493269 + 500 mg C10 | Cohort 2: 24 mg LY3493269 + 500 mg C10 | Cohort 3: 48 mg LY3493269 + 500 mg C10 | Cohort 4: 24 mg LY3493269 + 250 mg C10 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (6.6) | 44.9 (8.4) | 44.8 (9.1) | 44.9 (11.7) | 43.9 (8.1) | 43.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 8 | 8 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 8 | 8 | 8 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 8 | 8 | 8 | 8 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 8 | 8 | 8 | 8 | 8 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is an adverse event that results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.
Time Frame: Baseline through Day 43
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 8 mg LY3493269 + 500 mg C10: Participants received 8 milligrams (mg) LY3493269 + 500 mg permeation enhancer sodium caprate(C10) QD administered orally over 3 consecutive study days.
- 24 mg LY3493269 + 500 mg C10: Participants received 24 mg LY3493269 + 500 mg C10 QD administered orally over 3 consecutive study days.
- 48 mg LY3493269 + 500 mg C10: Participants received 48 mg LY3493269 + 500 mg C10 QD administered orally over 3 consecutive study days.
- 24 mg LY3493269 + 250 mg C10: Participants received 24 mg LY3493269 + 250 mg C10 QD administered orally over 3 consecutive study days.
Arm/Group | Placebo | 8 mg LY3493269 + 500 mg C10 | 24 mg LY3493269 + 500 mg C10 | 48 mg LY3493269 + 500 mg C10 | 24 mg LY3493269 + 250 mg C10
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3493269 From Day 1 and Day 3 Doses
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3493269.
  Note:
  1. 24 hour timepoint for Day 1 is the Day 2 pre-dose timepoint, which is the reason why Day 2 pre-dose is included in the timeframe.
  2. 24 hour timepoint for Day 3 is the Day 4 pre-dose timepoint, which is the reason why Day 4 pre-dose is included in the timeframe.
Time Frame: Day 1: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 2. 6, 8, 12 and Day 2 predose; Day 3: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hours post dose, Day 4, pre-dose
Population: All randomized participants received at least 1 full dose of LY3493269 and had evaluable PK sample. Participants may have been excluded from the PK summary statistics and statistical analysis if they had an adverse event of vomiting that occurred at or before 2 times median time to maximum observed drug Concentration (tmax)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | 8 mg LY3493269 + 500 mg C10 | 24 mg LY3493269 + 500 mg C10 | 48 mg LY3493269 + 500 mg C10 | 24 mg LY3493269 + 250 mg C10
Number analyzed (Participants) | 8 | 7 | 8 | 8
Nanograms per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 6 | 7 | 8 | 7
  Day 1 | 11.7 (176) | 39.9 (248) | 80.8 (359) | 68.2 (97)
  Day 3: number analyzed (Participants) | 8 | 6 | 7 | 8
  Day 3 | 17.7 (149) | 49.1 (449) | 41.9 (157) | 69.4 (263)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to 24 (AUC[0-24]) of LY3493269 From Day 1 and Day 3 Doses
Description: PK: Area Under the Concentration Versus Time Curve From Zero to 24 (AUC[0-24]) of LY3493269 From Day 1 and Day 3 Doses
  Note:
  1. 24 hour timepoint for Day 1 is the Day 2 pre-dose timepoint, which is the reason why Day 2 pre-dose is included in the timeframe.
  2. 24 hour timepoint for Day 3 is the Day 4 pre-dose timepoint, which is the reason why Day 4 pre-dose is included in the timeframe.
Time Frame: Day 1: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and Day 2 predose; Day 3: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hours post dose, Day 4, pre-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms hour per milliliter (ng*h/mL)
Arm/Group | 8 mg LY3493269 + 500 mg C10 | 24 mg LY3493269 + 500 mg C10 | 48 mg LY3493269 + 500 mg C10 | 24 mg LY3493269 + 250 mg C10
Number analyzed (Participants) | 8 | 7 | 8 | 8
Nanograms hour per milliliter (ng*h/mL)
  Day 1: number analyzed (Participants) | 6 | 7 | 8 | 7
  Day 1 | 170 (185) | 601 (310) | 1180 (381) | 1080 (104)
  Day 3: number analyzed (Participants) | 8 | 6 | 7 | 8
  Day 3 | 302 (139) | 868 (381) | 746 (156) | 1340 (276)

ADVERSE EVENTS:
Time Frame: Baseline Up To 43 Days
Arm/Group | Placebo | 8 mg LY3493269 + 500 mg C10 | 24 mg LY3493269 + 500 mg C10 | 48 mg LY3493269 + 500 mg C10 | 24 mg LY3493269 + 250 mg C10
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 7/8 | 8/8 | 7/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 8 mg LY3493269 + 500 mg C10 (N=8) | 24 mg LY3493269 + 500 mg C10 (N=8) | 48 mg LY3493269 + 500 mg C10 (N=8) | 24 mg LY3493269 + 250 mg C10 (N=8)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (4) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (10) | 2 (5) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 2 (3) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Catheter site erythema (General disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site phlebitis (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site erythema (General disorders) | 4 (4) | 3 (4) | 7 (9) | 5 (5) | 5 (6)
Medical device site injury (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Medical device site reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (5) | 0 (0) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT04498390/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT04498390/SAP_001.pdf